CLINICAL TRIAL: NCT05763004
Title: A Phase 1a/1b, First-in-human, Open-label, Non-randomized, Multicenter, Dose Escalation and Cohort Expansion Study to Evaluate the Safety, Tolerability, Efficacy, Immunogenicity, Pharmacokinetics, and Pharmacodynamics of IOS 1002 Administered Alone and in Combination with Pembrolizumab, a PD-1 Monoclonal Antibody in Advanced Solid Tumors
Brief Title: A Clinical Study to Evaluate the Safety, Tolerability and Efficacy of IOS-1002 Administered Alone and in Combination with Pembrolizumab, a PD-1 Monoclonal Antibody in Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ImmunOs Therapeutics AG (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IOS-1002-201; KEYNOTE-F49 / MK-3475-F49 (Other: Merck Sharp & Dohme, LLC)
Record Dates: First submitted 2023-01-09; First posted 2023-03-10 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-01

CONDITIONS: Solid Tumor, Adult
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IOS-1002 Monotherapy (Experimental)
  Interventions: Drug: IOS-1002
- IOS-1002 Combination Therapy with KEYTRUDA® (pembrolizumab) (Experimental)
  Interventions: Drug: IOS-1002 + KEYTRUDA® (pembrolizumab)

INTERVENTIONS:
Drug: IOS-1002 — monotherapy
  Arms: IOS-1002 Monotherapy
Drug: IOS-1002 + KEYTRUDA® (pembrolizumab) — combination therapy
  Arms: IOS-1002 Combination Therapy with KEYTRUDA® (pembrolizumab)

SUMMARY:
The goal of this clinical trial is to learn about IOS-1002 in patients with solid tumors.

The main questions it aims to answer are:

* To determine the safety and tolerability of various doses of IOS-1002 administered alone and/or in combination with KEYTRUDA® (pembrolizumab) in a single dose escalation scheme
* To determine the safety, tolerability and efficacy of a selected dose of IOS-1002 administered every 2 weeks alone and in combination with a PD-1 Antibody

The study will be conducted in 3 parts:

* Part A (Phase 1a, monotherapy and combination therapy dose escalation): IOS-1002 alone and IOS-1002 plus PD-1 mAb in patients with advanced solid tumors
* Part B (Phase 1b, monotherapy cohort expansion): IOS-1002 alone in patients with advanced solid tumors
* Part C (Phase 1b, combination therapy cohort expansion): IOS-1002 plus PD-1 mAb in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old at the time of Screening (signing the informed consent form [ICF]).
2. Histologically or cytologically confirmed advanced solid tumor (metastatic and/or unresectable) with measurable disease per RECIST v1.1:

   1. Malignancy that has relapsed or is refractory to, at least 1 standard treatment regimen in the advanced or metastatic setting, if such a therapy exists or for which the subjects who refuse or are ineligible for standard therapy.
   2. Subjects with lesions in a previously irradiated field as the sole site of measurable disease will be permitted to enrol provided the lesions have demonstrated clear progression and can be measured accurately.
3. For combination therapy dose-escalation: subjects who have undergone treatment with any agent specifically targeting checkpoint pathway inhibition (such as PD-1, PD-L1, PDL-2, LAG-3, or CTLA-4 antibody) for at least 3 months before disease progression and must have a gap of at least 4 weeks from the last treatment before receiving study treatment on Cycle 1 Day 1

   a. Subjects who experienced prior Grade 1 to 2 checkpoint therapy-related immune mediated AEs must have confirmed recovery from these events at the time of study entry, other than endocrinopathies treated with supplementation. Where applicable, these subjects must also have completed steroid tapers for treatment of these AEs by a minimum of 14 days prior to commencing treatment with study therapy. b) Eligibility of subjects with prior Grade ≥3 checkpoint therapy-related immune AEs, will be considered on a case-by-case basis after discussion with the Medical Monitor (eg, asymptomatic isolated Grade 3 lipase elevations without clinical or radiological features of pancreatitis will be permitted to enrol).
4. Adequate organ function at Screening
5. Willingness to provide consent to allow the acquisition of fresh tumor biopsy and/or existing formalin tissue sample
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1.

Exclusion Criteria:

1. Subjects with known or suspected CNS metastases, untreated CNS metastases, or with the CNS as the only site of disease are excluded. EXCEPTION: Subjects with controlled brain metastases will be allowed to enroll. Controlled brain metastases are defined as no radiographic progression for at least 4 weeks following radiation and/or surgical treatment (or 4 weeks of observation if no intervention is clinically indicated), and off steroids for at least 4 weeks prior to Screening, and no new or progressive neurological signs and symptoms.
2. Subjects with known carcinomatous meningitis.
3. Subjects with a prior malignancy except non-melanoma skin cancers, and in situ cancers such as: bladder, colon, cervical/dysplasia, melanoma, or breast. Subjects with other second malignancies diagnosed more than 2 years ago who have received therapy with curative intent with no evidence of disease during the interval who are considered by the Investigator to present a low risk for recurrence will be eligible.
4. Subjects with active, known, or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, euthyroid with a history of Grave's disease (subjects with suspected autoimmune thyroid disorders must be negative for thyroglobulin and thyroid peroxidase antibodies and thyroid-stimulating immunoglobulin prior to first dose of study treatment), psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
5. Subjects with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity, including subjects with pneumonitis.
6. Chronic Obstructive Pulmonary Disease (COPD) requiring recurrent steroids bursts or chronic steroids at doses greater than 10 mg/day of prednisone or the equivalent.
7. Uncontrolled or significant cardiovascular disease
8. Evidence of active infection ≤7 days prior to initiation of study treatment therapy (does not apply to viral infections that are presumed to be associated with the underlying tumor type required for study entry).
9. Evidence or history of active or latent tuberculosis infection including purified protein derivative recently converted to positive; chest x-ray with evidence of infectious infiltrate.
10. History of any chronic hepatitis
11. Known history of testing positive for HIV or known acquired immunodeficiency syndrome. Note: Testing for HIV must be performed at Screening.
12. Any anticancer therapy (eg, chemotherapy, biologics, vaccines, or hormonal treatment) including investigational drugs within 4 weeks prior to the first dose of study treatment administration, except for GnRH agonist therapy for subjects with prostate cancer and anticancer therapies with half-life of <4 weeks eg, prior use of EGFR TKI (completed at least two weeks prior to first dose of study treatment is acceptable).
13. Subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study treatment administration except for adrenal replacement steroid doses >10 mg daily prednisone equivalent in the absence of active autoimmune disease. Note: Treatment with a short course of steroids (<5 days) up to 7 days prior to initiating study treatment is permitted.
14. Use of non-oncology vaccines containing live virus for prevention of infectious diseases within 12 weeks prior to study treatment. The use of inactivated seasonal influenza vaccines eg, Fluzone® will be permitted on study without restriction.
15. Any major surgery within 4 weeks of study treatment administration. Subjects must have recovered from the effects of major surgery or significant traumatic injury at least 14 days before the first dose of study treatment.
16. Prior organ allograft.
17. Use of packed red blood cells (pRBC) or platelet transfusion within 2 weeks prior to the first dose of study treatment.
18. History of allergy to PD-1 mAb, significant drug allergy (such as anaphylaxis or hepatotoxicity) to prior anticancer immune modulating therapies (eg, checkpoint inhibitors, T-cell costimulatory antibodies).
19. All toxicities attributed to prior anticancer therapy other than alopecia and fatigue must have resolved to Grade 1 (NCI CTCAE v5.0) or baseline before administration of study treatment. Subjects with toxicities attributed to prior anticancer therapy which are not expected to resolve and result in long lasting sequelae, such as neuropathy after platinum-based therapy, are permitted to enroll.
20. Subjects with known HLA alloimmunization (not specifically tested for the trial)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
To determine the incidence of treatment emergent Adverse Events (Safety and Tolerability) of various doses of IOS-1002 administered alone and/or in combination with a PD-1 mAb in subjects with advanced solid tumors | From date of randomization until the date of first documented progression (end of study) or date of death from any cause, whichever came first, assessed up to 48 months
  Incidence of any Adverse Event DLTs AEs leading to study treatment discontinuationAEs leading to study discontinuation Abnormal laboratory parameters, vital signs, ECOG performance status, ECG results, and physical examination

SECONDARY OUTCOMES:
To investigate the preliminary antitumor activity of IOS-1002 and in combination with a PD-1 mAb | From date of randomization until the date of first documented progression (end of study) or date of death from any cause, whichever came first, assessed up to 48 months
  Investigator-assessed treatment response as defined and summarized by RECIST v1.1 and/or iRECIST
To characterize the PK of IOS-1002 alone and in combination with a PD-1 mAb | From date of randomization until the date of first documented progression (end of study) or date of death from any cause, whichever came first, assessed up to 48 months
  Concentrations of IOS-1002 in plasma
To characterize the immunogenicity of IOS-1002 alone and in combination with a PD-1 mAb | From date of randomization until the date of first documented progression (end of study) or date of death from any cause, whichever came first, assessed up to 48 months
  Number of subjects with ADA.
To characterize the immunogenicity of IOS-1002 | From date of randomization until the date of first documented progression (end of study) or date of death from any cause, whichever came first, assessed up to 48 months
  Percentage of subjects with ADA

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (5):
  - Monash Health Medical Center, Clayton
  - Austin Health / Cancer Clinical Trials Center, Heidelberg
  - Alfread Health, Melbourne
  - Peter MacCallum Cancer Center, Melbourne
  - Linear Clinical Research, Perth

IPD SHARING:
Plan to Share IPD: No